CLINICAL TRIAL: NCT03621033
Title: Methods of Colonic Transendoscopic Enteral Tubing: a Multicenter, Randomized Controlled Trial
Brief Title: Methods of Colonic Transendoscopic Enteral Tubing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TET-CN-170803
Record Dates: First submitted 2018-08-05; First posted 2018-08-08 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Colonic Transendoscopic Enteral Tubing
Keywords: transendoscopic enteral tubing; Microbiota Transplantation; transparent cap-assisted colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-transparent cap-assisted endoscopic intubation (Other): we do not use transparent cap-assisted endoscopic intubation.
  Interventions: Procedure: colonic transendoscopic enteral tubing
- transparent cap-assisted endoscopic intubation (Other): we use transparent cap-assisted endoscopic intubation in the second insertion.
  Interventions: Procedure: colonic transendoscopic enteral tubing

INTERVENTIONS:
Procedure: colonic transendoscopic enteral tubing — The procedure colonic transendoscopic enteral tubing is as follows:The TET tube was inserted into the ileocecal junction through the endoscopy channel at the first time of the cecal intubation after examination and evaluation of the whole colon. Then, the colonoscope was removed from the colon while the TET tube was maintained at the ileocecal junction. Then the endoscopy was inserted into the ileocecum again for affixing the TET tube to cecum with titanium clips.

SUMMARY:
Colonic transendoscopic enteral tubing (TET) is a novel, safe, convenient, and reliable way for fecal microbiota transplantation (FMT) and the whole-colon enema treatment. The aim of this study was to evaluate the methodology, efficiency, feasibility and safety of using transparent cap-assisted endoscopy for colon TET implantation.

DETAILED DESCRIPTION:
Our previous article has reported the method of colon TET. However, the investigators found that it was difficult to find the cavity because of the concentration of intestinal folds caused by the tube pulling after insertion of TET. It is well known that transparent cap-assisted colonoscopy is easier to flatten the semilunar folds and improve mucosal exposure. Here the investigators test the hypothesis that using transparent cap-assisted colonoscopy significantly decreases the second cecal intubation time which not only improve work efficiency, but also saves patients' anesthesia time and cost. Thus, the investigators design a prospective multicenter, randomized controlled trial. The aim of this study was to evaluate the methodology, efficiency, feasibility and safety of using transparent cap-assisted endoscopy for colon TET implantation.

ELIGIBILITY:
Inclusion Criteria:

* Diseases requiring total colonic administration and fecal microbiota transplantation.
* Patients and healthy Volunteers with the need to sample in deep colon .
* Age > 7 years.
* Must be able to Colonic Transendoscopic Enteral Tubing and no contraindication by endoscopic examination, consent colon TET implantation and not associated with severe intestinal lesions such as fistula, stenosis, complex perianal lesions, severe ileocecal or ascending colon lesions resulting in no proper site for titanium clip fixation.

Exclusion Criteria:

* Data was not recorded as required; Before and after implantation is not the same physician operation.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-05-10 (Estimated); Study Completion 2020-05-10 (Estimated)

PRIMARY OUTCOMES:
The second cecal intubation time | one day
  Record the time of colonoscopy from the anus to the ileal flap in the second insertion.

SECONDARY OUTCOMES:
Adverse events rate | All patients were followed up from date of intubation to one mouth after discharge
  Procedure-related and tube-related adverse events after procedure
TET success rate | one day
  The success rate of of the TET procedure
Maximum insertion pain score | one day
  Using numerical rating scale to evaluate maximum insertion pain score in non anesthesia. The digital grading method uses 0-10 to represent different levels of pain, with 0 as painless and 10 as severe. The classification standard of pain degree is: 0: no pain; 1-3: mild pain; 4-6: moderate pain; 7-10: severe pain.
Retention time of tube | three month
  Retention time of colonic transendoscopic enteral tubing
Tubing time | one day
  The tubing time is from advancement of the TET tube through the channel to the end of the tubing.
Titanium clip fixation time | one day
  Record the time required for fixing a titanium clip.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, MD; PhD, Study Chair — Nanjing Medical University
Locations (2):
- China (2):
  - Fmt-Dt-N-27/1350, Nanjing, Jiangsu
  - Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Peng Z, Xiang J, He Z, Zhang T, Xu L, Cui B, Li P, Huang G, Ji G, Nie Y, Wu K, Fan D, Zhang F. Colonic transendoscopic enteral tubing: A novel way of transplanting fecal microbiota. Endosc Int Open. 2016 Jun;4(6):E610-3. doi: 10.1055/s-0042-105205. Epub 2016 Apr 28. PMID 27556065
- [Result] Westwood DA, Alexakis N, Connor SJ. Transparent cap-assisted colonoscopy versus standard adult colonoscopy: a systematic review and meta-analysis. Dis Colon Rectum. 2012 Feb;55(2):218-25. doi: 10.1097/DCR.0b013e31823461ef. PMID 22228167